CLINICAL TRIAL: NCT04117035
Title: A Personalised Radiosurgery Procedure for People With Trigeminal Neuralgia to Improve Pain, Quality of Life and Reduce Complications - a Confidence in Concept Pilot Study (PROMOTION)
Brief Title: A Personalised Radiosurgery Procedure for People With Trigeminal Neuralgia to Improve Pain, Quality of Life and Reduce Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Jianhua Wu, Associate professor in Medical Statistics/Biostatistics, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 255351; 115658 (Other: University of Leeds)
Record Dates: First submitted 2019-09-18; First posted 2019-10-07 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Trigeminal Neuralgia; Multiple Sclerosis; Pain
Keywords: multiple sclerosis; trigeminal neuralgia; Pain; Quality of life
MeSH Terms: conditions — Trigeminal Neuralgia; Multiple Sclerosis; Pain | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: single-blinded randomised control pilot study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): Standard care
  Interventions: Procedure: GKRS standard care
- Intervention (Experimental)
  Interventions: Procedure: Gamma Knife Radiosurgery (GKRS) personalised procedure

INTERVENTIONS:
Procedure: Gamma Knife Radiosurgery (GKRS) personalised procedure — Personalised GKRS treatment
  Arms: Intervention
Procedure: GKRS standard care — Standard GKRS treatment
  Arms: Control arm

SUMMARY:
The aim of this study is to evaluate prospectively the feasibility and impact of personalised gamma knife radiosurgery treatment protocol versus current standard protocol for people with idiopathic or Multiple Sclerosis-related Trigeminal Neurolgia (MS related TN) on effectiveness in pain relief, the development of morbidity and quality of life.

Patients with TN or MS-related TN are referred to the National Centre for Stereotactic Radiosurgery in Sheffield for clinical consultation, and will undergo gamma knife radiosurgery (GNRS) for treating trigeminal neuralgia if eligible. The GKRS treatment is provided as a standard National Health Service (NHS) routine care. The current procedure has been proven to be safe and effectiveness in reducing the pain caused by TN. The current GKRS treatment protocol performs the treatment on the trigeminal nerve close to the brainstem, which might result in higher complication rate (mainly facial numbness). This study will conduct a pilot randomised controlled trial to evaluate an alternative treatment protocol, which will perform the GKRS treatment at the retrogasserian zone (further away from the brainstem). This treatment protocol has been widely used in Europe and USA, and is safe and effective. Most studies adopting this protocol have shown less complication rate after treatment.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a condition of excruciating facial pain characterized by brief, repeated, electric shock-like pains. Like idiopathic TN, people with multiple sclerosis (MS) related TN (PwMSTN) often suffer from episodic facial pain (often excruciating) that may be related to demyelination of the trigeminal pathways. It is estimated that people with multiple sclerosis (PwMS) are 20 times more likely to present with TN symptoms than non-MS people and a recent review estimated that 4-8% of PwMS have TN. Patients with TN or MS-related TN who no longer respond to treatment often opt for non-invasive gamma knife radiosurgery (GKRS), with variable outcomes. Factors, such as patient characteristics, target treatment location and radiation dosage, could affect the efficacy of pain relief and result in post-surgical morbidity. There is no consensus of the best GKRS target treatment location or the optimal radiation dosage for GKRS treatment among centers, this results in great variability across centers in patient outcomes of pain control and morbidity. This prospective surgical pilot study will recruit PwTN and PwMS-related TN from the National Center for Stereotactic Radiosurgery, Sheffield, to evaluate the impact of a personalized GKRS treatment protocol on safety, efficacy (pain control) and morbidity. The personalized procedure will target the treatment location on trigeminal nerve further away from the brain stem as compared to the current standard treatment location that is closer to the brain stem. The personalized procedure may reduce the radiation dose to the brain stem and then reduce the adverse effects of the treatment. The recruited PwTN and PwMS-related TN will be randomly allocated to either the personalized GKRS treatment protocol group or the standard GKRS treatment protocol group. The efficacy in pain relief and morbidity will be evaluated between the treatment groups at 6 months and 12 months post-surgery.

This study does not have main ethical, legal issues. The GKRS treatment is provided as routine NHS care, and the study will only alter the treatment location for those patients who would normally go through the standardtreatment protocol. Therefor there will be no management issues.

Information collected during this study will be kept confidential. All data collected for this study will be kept safely and securely on secure NHS computer server and paper records at the clinic. All data will be handled strictly according to the University of Leeds privacy notice for research participants

ELIGIBILITY:
Inclusion Criteria:

1. Subject has idiopathic TN or MS-related TN.
2. Subject is available for follow up.

4. Subject can understand the informed consent form in English. 5. Age over 18 years at the time of signing the Informed Consent Form 6. Have been treatment planned to receive GKRS treatment

Exclusion Criteria:

Patients who:

1. Have no capacity to complete written informed consent
2. Do not understand English
3. Repeat GKRS treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Barrow Neurological Institute (BNI) pain measure | 6 MONTHS
  BNI Pain Scale (BNI-PS), 5-level categories (scale range: 1-5)
Barrow Neurological Institute (BNI) numbness measure | 6 MONTHS
  BNI Numbness Scale (BNI-NS), 5-level categories (scale range: 1-5)

SECONDARY OUTCOMES:
Current medication and dosage | 12 MONTHS
Vision complications | 12 MONTHS
  Recorded as adverse events such as blurred vision, double vision, or water eyes
Motor impairment | 12 MONTHS
  Assessed through a battery of test with a performance score (range: 1-100)
Cognitive impairment | 12 MONTHS
  Assessed through a battery of test with a performance score (range: 1-100)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wu, PhD, Principal Investigator — University of Leeds
Locations (1):
- Sheffield royal hallamshire hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No